CLINICAL TRIAL: NCT01813123
Title: A Web-Based Intervention to Prevent Drug Abuse Among Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Traci M. Schwinn, Associate Research Scientist, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAJ3409; R01DA031782 (NIH)
Record Dates: First submitted 2013-03-08; First posted 2013-03-18 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Drug Abuse Prevention
Keywords: gender-specific; web-based; drug abuse; prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): RealTeen
  Interventions: Behavioral: RealTeen

INTERVENTIONS:
Behavioral: RealTeen — A web-based, gender-specific program intended improve girls' cognitive and behavioral skills. Each of the 9 sessions requires approximately 20 minutes. After initial intervention, girls will receive two annual booster sessions (i.e., a 20-minute review of previously learned material indexed to new age).
  Arms: Intervention

SUMMARY:
This study is designed to develop and test a gender-specific, web-based drug abuse prevention program. Study participants will be adolescent girls aged 13 and 14 years who will complete all measures online. Randomly assigned girls will also interact online with a skills-based program and subsequent annual booster sessions.

The study's primary hypothesis is that rates of 30-day alcohol and drug use will be lower among girls assigned to receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* resident of USA
* speaks English
* have private computer with Internet

Exclusion Criteria:

-

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 788 (Actual)
Dates: Start 2013-03; Primary Completion 2017-07 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
30-day alcohol and drug use | Up to 3 years
  Measures will ask girls to report, for the past 30 days, the number of: drinks of alcohol consumed, cigarettes smoked, puffs of marijuana, and times they consumed four or more drinks within 2 hours. Girls will also report past 30-day use of: inhalants, ecstasy, club drugs, prescription drugs for recreational use, heroin, and hallucinogens.

CONTACTS AND LOCATIONS:
Overall Officials: Traci M Schwinn, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Social Work, New York, New York, United States